CLINICAL TRIAL: NCT06074471
Title: Motor Sparing Supraclavicular Brachial Plexus Block (MS-SCBPB): A Randomized Controlled Trial
Brief Title: Motor Sparing Supraclavicular Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nagy Malak , MD, Lecturer of anesthesia ,SICU and pain, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-267-2023
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia; Regional Anesthesia Morbidity
Keywords: Motor sparing; SCBP block; Upper limb operations
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Drugs used (bupivacaine-lidocaine-Dexamethazone) Rescue analgesic is morphine
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS-SCBPB Group (n=22) (Experimental): receive ultrasound-guided supraclavicular brachial plexus block with total volume 20 mL bupivacaine (concentration 0.20%) "9 ml Bupivacaine+9ml lignocaine +2ml Dexamethasone 8mg "
  Interventions: Procedure: ultrasound guided supraclavicular brachial plexus block
- SCBPB Group (n=22): (Active Comparator): receive ultrasound-guided supraclavicular brachial plexus block with total volume 20 mL bupivacaine (concentration 0.5%) "18 ml Bupivacaine+2ml Dexamethasone 8mg"
  Interventions: Procedure: ultrasound guided supraclavicular brachial plexus block

INTERVENTIONS:
Procedure: ultrasound guided supraclavicular brachial plexus block — Block will be performed in semi-sitting position with head tilted to the opposite side of injection site. linear probe (4-12MHz) (Mindray Digital Ultrasonic Model DP-10 "SN 6N-49005130" 2014-09. SHENZHEN MINDRAY BIO-MEDICAL ELECTRONICS CO.LTD) will be placed parallel to the clavicle in the supraclavicular fossa visualizing the subclavian artery is seen beating above the first rib. A volume of 2 mL lignocaine 2% will be infiltrated subcutaneous before the block. A 20-gauge needle will be advanced in plane aiming to the corner pocket towards the deeper portion of the brachial plexus at the angle between the first rib and the subclavian artery, 10 mL of drug will be injected. Then, the needle will be retracted and advanced at a shallower angle, aiming toward the superficial plexus after negative aspiration another 10 ml will be injected, total drug injected 20 ml (18 mL of drug will be injected with addition to 8mg dexamethasone (2ml))
  Other Names: Drugs used (bupivacaine and dexamethazone)

SUMMARY:
This study aims to compare MS-SCBPB and SCBPB in the duration of postoperative analgesia, time to first analgesic request (VAS ≥40 mm), pain scores, motor power, and side effects.

DETAILED DESCRIPTION:
On arrival of the patients to regional anesthesia room, patients will be secured with 20-gauge intravenous cannula. Monitoring will include ECG, non-invasive arterial blood pressure, and pulse oximetry (SpO2).

Before receiving supraclavicular brachial plexus block, patients will be randomly assigned into one of the two study groups:

MS-SCBPB Group (n=22): this group will receive ultrasound-guided supraclavicular brachial plexus block with total volume 20 mL bupivacaine 0.20% and 8 mg dexamethasone.

SCBPB Group (n=22): this group will receive ultrasound-guided supraclavicular brachial plexus block with total volume 20 mL bupivacaine 0.5% and 8 mg dexamethasone.

Another doctor not involved in the block procedure will evaluate the patients postoperative.

Technique of SCBPB:

The technique of ultrasound-guided supraclavicular brachial plexus block will be performed with the patient in semi-sitting position with head tilted to the opposite side of injection site. A linear ultrasound probe (4-12MHz) will be placed parallel to the clavicle in the supraclavicular fossa visualizing the subclavian artery is seen beating above the first rib. A volume of 2 mL lignocaine 2% will be infiltrated subcutaneous before the block. A 20-gauge needle will be advanced in plane under direct vision aiming to the corner pocket towards the deeper portion of the brachial plexus at the angle between the first rib and the subclavian artery, a total of 10 mL of drug will be injected, aspirating every 5 ml. Then, the needle will be retracted and advanced at a shallower angle, aiming toward the superficial brachial plexus after negative aspiration, 10 mL of drug will be injected, aspirating every 5 ml.

Block assessment:

Time needed for surgical block: the time interval from the end of ultrasound guided supraclavicular brachial plexus block injection till achievement surgical anesthesia

Assessment of surgical anesthesia using a 3-point score:

Extent of sensory block:

In all four nerves: hypothenar eminence (ulnar nerve), thenar eminence (median nerve), dorsum of hand (radial nerve), and lateral aspect of the forearm (musculocutaneous nerve) 0 = loss of sensation to light touch, 1 = loss of sensation to pinprick, 2 = normal sensation

Extent of motor block:

In all four nerves: thumb adduction (ulnar nerve), thumb opposition (median nerve), thumb abduction (radial nerve), and flexion of the elbow in supination and pronation (musculocutaneous nerve) 0 = no movement, 1 = paresis, 2 = normal movement Interpretation : Block success for surgical anesthesia is defined as the achievement of sensory and or motor scores of 1 or less at 5, 10, 15, 20, and 30 minutes post-injection.

Intraoperative Care:

An anesthesiologist blinded to group allocation will be attending for monitored anesthesia care with a safe conscious sedation intraoperatively, titrated to patient comfort using low intravenous doses of midazolam (1-3mg), fentanyl (1-2 μg/kg), and/or Propofol (25-75 μg/kg/min). In the event of failed block, it will be managed with either local anesthetic supplementation at the corresponding spared nerve or converted to general anesthesia.

Postoperatively, all patients will receive 1 g paracetamol every 6 h and 30 mg ketorolac every 12 h. Intravenous morphine titration will be carried out at patient wake-up to achieve pain control (Using visual analogue scale (VAS) for pain assessment from 0 the Best to 10 the worst) by an attending anesthesiologist blinded to group allocation. Patients with a VAS score of ≥ 4 and patients who will request rescue analgesia will be treated with IV morphine in 2 mg increments every 4 hours with upper limit for the total administered dose (maximum 20 mg per day). If the patient appeared sedated (Ramsay sedation scale > 2), and/or severe morphine-related side effects are encountered including respiratory depression (Spo2 < 95% and/or RR < 12 breaths/min), allergic reaction, hypotension, or severe pruritus, morphine titration will be stopped and the patient will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for upper limb surgeries under supraclavicular brachial plexus block
* American Society of Anesthesiologists (ASA) status I and III
* between ages of 18 and 60 years

Exclusion Criteria:

* Bleeding disorders with INR > 1.5 and/or platelets < 100,000/mm3
* infection at the injection site
* Allergy to local anesthetics
* Severe cardiopulmonary disease (≥ASA IV)
* Diabetic or other neuropathies
* Motor disorders
* Patients receiving opioids for chronic analgesic therapy
* Inability to comprehend visual analogue scale (VAS).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Duration of motor blockade | 24 hours
  Duration of motor blockade

SECONDARY OUTCOMES:
Time needed for surgical block: | 24 hours
  the time interval between the injection of the study medication till surgical anesthesia.
Time needed for complete recovery from sensory and motor block at 2, 4, 6, 12, 18, and 24 hours postoperatively. | 24 hours
  Time needed for complete recovery from sensory and motor block at 2, 4, 6, 12, 18, and 24 hours postoperatively.
Time to first analgesic request | 24 hours
  Time to first analgesic request Using Visual analogue scale (VAS) for pain assessment from 0 the Best to 10 the worst) ...rescue analgesic given if VAS >4
Visual analogue scale (VAS) | 24 hours
  Visual analogue pain score for pain assessment from 0 the Best to 10 the worst) at 2, 4, 6, 12, 18, and 24 hours postoperatively.
Total morphine requirements | 24 hours
  Total morphine requirements 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university Hospitals. kasralainy, Cairo, Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No